CLINICAL TRIAL: NCT04972500
Title: The Influence of Fasting on Selected Hemodynamic Parameters Measured in a Non-invasive Way
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Clinical Professor, Head of Department of Anaesthesiology and Intensive Care, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREOP2
Record Dates: First submitted 2021-07-09; First posted 2021-07-22 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Perioperative Complication; Hemodynamic Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-op (Experimental): Nutricia Pre-op, 400 milliliters, per os
  Interventions: Dietary Supplement: Nutricia Pre-op, 400 milliliters, per os
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Nutricia Pre-op, 400 milliliters, per os — After 10 hours of fasting participants will receive per os 400 milliliters of Nutricia Pre-op
  Arms: Pre-op

SUMMARY:
Preoperative fasting is considered to be refraining from taking meals for at least 6 hours and clear fluids for at least 2 hours before anesthesia. On the one hand, it is a procedure that reduces the risk of aspiration of chyme and the occurrence of Mendelson's syndrome, and on the other hand, it is one of the causes of water and carbohydrate disturbances in patients undergoing general anesthesia. Most of them experience some degree of dehydration in the preoperative period. It is associated with a worse prognosis. Due to the negative impact of fasting on homeostasis, as well as significant changes in heart rate in participants in the previous study, we decided to measure the hemodynamic parameters during fasting. The development of impedance cardiography techniques enables the measurement of these parameters by a non-invasive method.

After obtaining the participant's written consent to participate in the study, the first measurement of body weight, blood pressure using a non-invasive method and hemodynamic parameters using a non-invasive impedance cardiography method using the Niccomo ™ device (Medizinische Messtechnik GmbH) will be performed in the evening. The subject will then be asked to refrain from food for at least 10 hours and fluid for 6 hours before the next measurement. The next morning, another measurement will be made and the participant will be randomly assigned to one of two groups: subjects in the first group will be asked to refrain from eating and drinking for another 2 hours, while subjects in the second group per os will receive 400 milliliters of PreOp® (Nutricia ™ preparation intended for preoperative dietary management in surgical patients, containing carbohydrates and electrolytes). After another two hours, the third measurement of the tested parameters will be performed. The obtained results will be subjected to statistical analysis consisting in comparing the values of hemodynamic parameters between the studied groups at appropriate measurement points.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) general condition assessment 1 or 2

Exclusion Criteria:

* Chronic kidney disease
* Circulatory failure
* Lung diseases
* Diseases of the heart valves
* History of hypoglycaemic episodes or any carbohydrate disturbance.
* Height less than 120 cm or greater than 230 cm
* Body weight less than 30 kg or greater than 155 kg.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac index (CI) | Changes form baseline after 10 hours of fasting and after 2 hours of pre-op administration
  Cardiac index will be measured non-invasively with Niccomo™(Medizinische Messtechnik GmbH) device.
  Cardiac index will be measured in l/min/m^2 (liters per minute per square meter).
Changes in systemic vascular resistance index (SVRI) | Changes form baseline after 10 hours of fasting and after 2 hours of pre-op administration
  Systemic vascular resistance index will be measured non-invasively with Niccomo™(Medizinische Messtechnik GmbH) device.
  Systemic vascular resistance index will be measured in dyn*s*cm^-5*m^2 (dyne multiply by second multiply by centimeters to the power of minus 5 multiply by square meter)
Changes in stroke volume (SV) | Changes form baseline after 10 hours of fasting and after 2 hours of pre-op administration
  Stroke volume will be measured non-invasively with Niccomo™(Medizinische Messtechnik GmbH) device.
  Stroke volume will be measured in mL (milliliters).
Changes in heart rate (HR) | Changes form baseline after 10 hours of fasting and after 2 hours of pre-op administration
  Heart rate will be measured non-invasively with Niccomo™(Medizinische Messtechnik GmbH) device.
  Heart rate will be measured in 1/min (beats per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Owczuk, Prof., Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk - Departament of Anesthesiology and Intensive Care, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No